CLINICAL TRIAL: NCT06565247
Title: Evaluation of PSMA-PET and mpMRI in High-risk Prostate Cancer - Using Histopathologic Validation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Västerbotten (Other Government)
Collaborators: Umeå University (Other); Region Skane (Other); Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAMP2; CIV-23-04-042756 (Other: Swedish Medical Products Agency); 2022-501892-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-surgical imaging of high-risk prostate cancer using [18F]PSMA-PET/mpMRI or mpMRI (Experimental): One-time pre-surgical imaging using [18F]PSMA-PET/mpMRI (at Umea University Hosptial) or mpMRI (at Skåne University Hospital)
  Interventions: Drug: [18F]PSMA-PET; Device: MRI sequences optimized for prostate cancer examinations

INTERVENTIONS:
Drug: [18F]PSMA-PET — Pre-surgical imaging using [18F]PSMA-PET at Umea University Hospital, 3.5 MBq/kg, i.v. injection.
Device: MRI sequences optimized for prostate cancer examinations — T2-WI, T1-WI, DCE and DWI at Umea University Hospital and at Skåne University Hospital

SUMMARY:
In this trial the connection between image properties (mpMRI and PSMA-PET) and tissue properties (molecular and histopathology) will be investigated in order to improve diagnostics and image-based treatment guidance of prostate cancer.

DETAILED DESCRIPTION:
Open, non-randomized, prospective multi-center trial, with consecutive recruiting, between Skåne University hospital and Umeå University Hospital.

High-risk prostate cancer patients referred for radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer planned to be treated with radical prostatectomy
2. PSMA-PET/CT conducted as part of the clinical management for the existing prostate cancer.
3. ≥4 weeks since last biopsy of the prostate
4. One or more of the following criteria

   1. cT3, or high suspicion of extra prostatic growth on mpMRI
   2. Gleason score ≥8
   3. PSA 20-49 ng/ml
5. >18 years
6. Given a written consent to participate in the trial

Exclusion Criteria:

1. Non-MR-safe implants or another contraindication to MRI or PET
2. Claustrophobia
3. Unfit for MRI or PET/MRI examination for any other reason, e.g., back pain
4. WHO PS >1
5. Patients treated with neoadjuvant/concomitant anti-testosterone treatment (surgical or medical castration or anti-androgens)
6. TUR-P within 6 months
7. Metastatic disease in skeleton, parenchymal organs, or lymph nodes outside the pelvis.
8. Patients with previous diagnosis of other malignant disease. Exceptions could be made for basal cell carcinoma of the skin or progression free survival at least 10 years after any previous tumour.
9. Creatinine clearance < 30ml/min (acc. to http://www.fass.se/LIF/produktfakta-/kreatinin.jsp)
10. Tinnitus or severe hearing loss

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of PSMA-PET and mpMRI for identification and delineation of intraprostatic lesions | Pre-surgical imaging 1-6 weeks before surgery vs. post-surgery histopathology as performed within 1-4 weeks for normal clinical work-up. Within the 5-year time frame of the study, analyses will be complemented with detailed study specific histopathology
  Spatially defined aggressive PC lesions, or subparts of lesion, identified and defined using PSMA-PET and/or mpMRI compared to histopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Thellenberg Karlsson, MD, PhD, Principal Investigator — Region Västerbotten
Locations (2):
- Sweden (2):
  - Region Skåne, Malmo
  - Region Västerbotten, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Trial data that are possible to de-identify (anonymize) will be made available to other research groups through an open repository such as https://zenodo.org or equivalent. Shared data will not be directly traceable to an individual participant.
Supporting Information: Study Protocol
Time Frame: Study protocol and anonymized data will be made available after study closure.
Access Criteria: Study protocol will be publicly available. Anonymized data will be accessible by request.